CLINICAL TRIAL: NCT03333109
Title: A 12-week Double-blind, Randomized, Multi-center Study Comparing the Efficacy and Safety of Once Monthly Subcutaneous AMG 334 Against Placebo in Adult Episodic Migraine Patients (EMPOwER)
Brief Title: Study of Efficacy and Safety of AMG 334 in Adult Episodic Migraine Patients
Acronym: EMPOwER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAMG334A2302
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2021-03-09 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Episodic Migraine
Keywords: AMG334; erenumab; episodic migraine; headache; CGRP; Calcitonin Gene-related; migraine; adult
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AMG334 70 mg (Experimental): AMG334 70 mg: one pre-filled syringe containing 70 mg of erenumab plus one pre-filled syringe of identical placebo administered subcutaneous every 28 days
  Interventions: Biological: Erenumab
- AMG334 140 mg (Experimental): AMG334 140 mg: two pre-filled syringe containing 70 mg each of erenumab administered subcutaneous every 28 days
  Interventions: Biological: Erenumab
- Placebo (Placebo Comparator): Two pre-filled syringes containing placebo identical in appearance to erenumab
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Erenumab — 70 mg/mL pre-filled syringe administered subcutaneously
  Other Names: AMG334
  Arms: AMG334 140 mg; AMG334 70 mg
Other: Placebo — Matching placebo in pre-filled syringe administered subcutaneously
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy and safety of AMG334 in adult patients with episodic migraine

DETAILED DESCRIPTION:
This study used a single-cohort, 3-treatment arm, randomized, double-blind study design in adult patients with episodic migraine. The subjects were randomized to receive either erenumab or placebo in a 2:3:3 ratio (erenumab 140 mg: erenumab 70 mg: placebo). A screening period of 2 weeks was used to assess initial eligibility, followed by a 4-week baseline period. After randomization/Day 1, visits occurred at four week intervals until Week 12, which was the End of Treatment. The final visit, Last Patient Last Visit was a Safety Follow-Up visit, which occurred 12 weeks later, at Week 24.

ELIGIBILITY:
Key inclusion criteria:

1. Documented history of migraine in the 12 months prior to screening
2. 4-14 days per month of migraine symptoms
3. >=80% diary compliance during the Baseline period

Key exclusion criteria:

1. >50 years old at migraine onset
2. Pregnant or nursing
3. History of cluster or hemiplegic headache
4. Evidence of seizure or major psychiatric disorder
5. Score of 19 or higher on the BDI
6. Active chronic pain syndrome
7. Cardiac or hepatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Córdoba
- India (21):
  - Novartis Investigative Site, Guntur, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Thiruvananthapuram, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Belagavi
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
- Lebanon (2):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
- Malaysia (5):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuala Lumpur, MYS
  - Novartis Investigative Site, Seberang Jaya, Pulau Pinang
  - Novartis Investigative Site, Sungai Buloh, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Chihuahua City
- Philippines (3):
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon City
- Novartis Investigative Site, Singapore, Singapore
- South Korea (9):
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Daejeon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, KOR
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Taiwan (6):
  - Novartis Investigative Site, Chiayi City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taichung County
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (4):
  - Novartis Investigative Site, Bangkok, THA
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Vietnam (2):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wang SJ, Roxas AA, Saravia B, Kim BK, Chowdhury D, Riachi NJ, Tai MS, Tanprawate S, Tran TN, Zhao YJ, Su W, Wen S, Mondal S, Ecochard L, Arkuszewski M. Effect of Erenumab on Patient-Reported Outcomes in Episodic Migraine in Asia, the Middle East, and Latin America: Results From the EMPOwER Study. Neurol Clin Pract. 2026 Apr;16(2):e200565. doi: 10.1212/CPJ.0000000000200565. Epub 2026 Feb 2. PMID 41641373
- [Derived] Lampl C, Kraus V, Lehner K, Loop B, Chehrenama M, Maczynska Z, Ritter S, Klatt J, Snellman J. Safety and tolerability of erenumab in individuals with episodic or chronic migraine across age groups: a pooled analysis of placebo-controlled trials. J Headache Pain. 2022 Aug 18;23(1):104. doi: 10.1186/s10194-022-01470-4. PMID 35978286
- [Derived] Wang SJ, Roxas AA Jr, Saravia B, Kim BK, Chowdhury D, Riachi N, Tai MS, Tanprawate S, Ngoc TT, Zhao YJ, Mikol DD, Pandhi S, Wen S, Mondal S, Tenenbaum N, Hours-Zesiger P. Randomised, controlled trial of erenumab for the prevention of episodic migraine in patients from Asia, the Middle East, and Latin America: The EMPOwER study. Cephalalgia. 2021 Nov;41(13):1285-1297. doi: 10.1177/03331024211024160. Epub 2021 Jun 25. PMID 34171973
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=731

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Treatment Period (DBTP)
Arm/Group | AMG334 70 mg | AMG334 140 mg | Placebo
Started | 338 | 224 | 338
Full Analysis Set (All participants who started the study medication and completed at least one post-baseline efficacy measurement) | 329 | 219 | 330
Safety Analysis Set (Safety analysis set consisted of all randomized subjects who received at least one dose of investigational product and were analyzed based on the actual treatment received) | 335 | 224 | 335
Completed | 321 | 218 | 326
Not Completed | 17 | 6 | 12
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 4 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 6 | 5
Not completed — Randomized but not treated | 3 | 0 | 3
Period: Safety Follow-up Period
Arm/Group | AMG334 70 mg | AMG334 140 mg | Placebo
Started | 324 (Subjects discontinued from DBTP and still entered the safety follow-up.) | 218 | 328 (Subjects discontinued from DBTP and still entered the safety follow-up.)
Completed | 311 | 214 | 315
Not Completed | 13 | 4 | 13
Not completed — Lost to Follow-up | 6 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 2 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG334 70 mg | AMG334 140 mg | Placebo | Total
Number analyzed (Participants) | 338 | 224 | 338 | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (10.0) | 37.1 (9.6) | 38.0 (10.1) | 37.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 184 | 281 | 737
  Male | 66 | 40 | 57 | 163
Race/Ethnicity, Customized [Number; unit: participants] — If multiple races were reported for a participant, the participant was categorized as multiple and in each selected race category
  participants
    White | 58 | 35 | 60 | 153
    Black or African American | 1 | 0 | 0 | 1
    Asian | 278 | 184 | 269 | 731
    American Indian or Alaska Native | 1 | 0 | 1 | 2
    Multiple | 9 | 8 | 5 | 22
    Other | 9 | 13 | 13 | 35
Monthly Migraine Days at Baseline [Mean (Standard Deviation); unit: Migraine days/month] — A migraine day was defined as any calendar day in which the subject experienced a qualified migraine headache defined as a migraine with or without aura, lasting for ≥ 30 minutes, and meeting at least one of the following criteria:
  1. ≥ 2 of the following pain features: unilateral, throbbing, moderate to severe or exacerbated with exercise/physical activity
  2. ≥ 1 of the following associated symptoms: nausea and/or vomiting, photophobia and phonophobia Population: This analysis is based on the data available for computing the monthly migraine days, according to pre-specified algorithm
  Migraine days/month
    number analyzed (Participants) | 337 | 224 | 338 | 899
    (all) | 8.09 (2.62) | 8.27 (3.14) | 8.35 (2.76) | 8.23 (2.81)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days at the Last Month (Month 3) of the Double-blind Treatment Period (DBTP)
Description: A migraine day was defined as any calendar day in which the subject experienced a qualified migraine headache defined as a migraine with or without aura, lasting for ≥ 30 minutes, and meeting at least one of the following criteria:
  1. ≥ 2 of the following pain features: unilateral, throbbing, moderate to severe or exacerbated with exercise/physical activity
  2. ≥ 1 of the following associated symptoms: nausea and/or vomiting, photophobia and phonophobia
Time Frame: Baseline up to Month 3
Population: Full analysis set
Measure: Mean (Standard Error); unit: Migraine days/month
Arm/Group | AMG334 70 mg | AMG334 140 mg | Placebo
Number analyzed (Participants) | 329 | 219 | 330
Migraine days/month | -4.20 (0.25) | -4.79 (0.30) | -3.10 (0.25)
Statistical Analysis 1: Comparison: AMG334 70 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-1.77 to -0.42], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: AMG334 140 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -1.69, 95% CI 2-sided [-2.45 to -0.93], Standard Error of Mean 0.39

2. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Monthly Migraine Days at Month 3
Description: Achievement of at least a 50% reduction from baseline in monthly migraine days at Month 3. A migraine day was defined as any calendar day in which the subject experienced a qualified migraine headache defined as a migraine with or without aura, lasting for ≥ 30 minutes, and meeting at least one of the following criteria:
  1. ≥ 2 of the following pain features: unilateral, throbbing, moderate to severe or exacerbated with exercise/physical activity
  2. ≥ 1 of the following associated symptoms: nausea and/or vomiting, photophobia and phonophobia
Time Frame: Baseline and at Month 3
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | AMG334 70 mg | AMG334 140 mg | Placebo
Number analyzed (Participants) | 329 | 219 | 330
percentage of participants | 55.3 | 63.9 | 44.8
Statistical Analysis 1: Comparison: AMG334 70 mg vs Placebo; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Haenszel (CMH) test adjusted for stratification factor after missing data were imputed as non-response (NRI); Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.12 to 2.07]
Statistical Analysis 2: Comparison: AMG334 140 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Haenszel (CMH) test adjusted for stratification factor after missing data were imputed as non-response (NRI); Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.55 to 3.15]

3. Secondary Outcome: Change From Baseline in Acute Migraine-specific Medication Treatment Days at Month 3
Description: Number of days on which acute migraine-specific medications were used were recorded in eDiary between each monthly IP dose. Migraine-Specific medications include two categories of medications: triptan-based migraine medications and ergotamine-based migraine medications. Monthly migraine-specific medication use at baseline is the number of migraine-specific medication treatment days in the baseline period.
Time Frame: Baseline up to Month 3
Population: Analysis set included participants with at least one acute migraine-specific medication use during baseline
Measure: Mean (Standard Error); unit: Migraine days/month
Arm/Group | AMG334 70 mg | AMG334 140 mg | Placebo
Number analyzed (Participants) | 123 | 80 | 127
Migraine days/month | -1.84 (0.26) | -2.39 (0.33) | -0.49 (0.26)
Statistical Analysis 1: Comparison: AMG334 70 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-2.07 to -0.64], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: AMG334 140 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.90, 95% CI 2-sided [-2.71 to -1.09], Standard Error of Mean 0.41

4. Secondary Outcome: Change From Baseline in Headache Impact Scores as Measured by the Headache Impact Test (HIT-6) at Month 3
Description: The HIT-6 is a short-form self-administered questionnaire based on the internet-HIT question pool. The HIT-6 was developed as a global measure of adverse headache impact to assess headache severity in the previous month and change in a patient's clinical status over a short period of time. Six items assess the frequency of pain severity, headaches limiting daily activity (household, work, school, and social). Each of the 6 questions is responded to using 1 of 5 response categories: "never," "rarely," "sometimes," "very often," or "always." For each HIT-6 item, 6, 8, 10, 11, or 13 points, respectively, are assigned to the response provided. These points were summed to produce a total HIT-6 score that ranges from 36 to 78. Scores were categorized into 4 grades, representing little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78) due to headache. Lower values represent better outcomes, therefore negative change denotes improveme
Time Frame: Baseline up to Month 3
Population: Analysis included participants with a non-missing value at the corresponding time point of interest
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | AMG334 70 mg | AMG334 140 mg | Placebo
Number analyzed (Participants) | 296 | 200 | 308
scores on a scale | -8.39 (0.45) | -9.34 (0.54) | -6.62 (0.44)
Statistical Analysis 1: Comparison: AMG334 70 mg vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -1.77, 95% CI 2-sided [-2.99 to -0.56], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: AMG334 140 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.71, 95% CI 2-sided [-4.07 to -1.36], Standard Error of Mean 0.69

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 12 weeks post treatment, up to maximum duration of 28 weeks
Groups:
- AMG 334 70mg: AMG334 70 mg: one pre-filled syringe containing 70 mg of erenumab plus one pre-filled syringe of identical placebo administered subcutaneous every 28 days
- AMG 334 140mg: AMG334 140 mg: two pre-filled syringe containing 70 mg each of erenumab administered subcutaneous every 28 days
Arm/Group | AMG 334 70mg | AMG 334 140mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/335 | 0/224 | 0/335
Serious Adverse Events (participants affected / at risk) | 10/335 | 0/224 | 5/335
Other Adverse Events (participants affected / at risk) | 83/335 | 58/224 | 85/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 334 70mg (N=335) | AMG 334 140mg (N=224) | Placebo (N=335)
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 2 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 334 70mg (N=335) | AMG 334 140mg (N=224) | Placebo (N=335)
Constipation (Gastrointestinal disorders) | 20 | 12 | 10
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 6
Gastritis (Gastrointestinal disorders) | 0 | 1 | 4
Nausea (Gastrointestinal disorders) | 3 | 2 | 6
Fatigue (General disorders) | 4 | 3 | 0
Injection site erythema (General disorders) | 4 | 1 | 8
Injection site pain (General disorders) | 4 | 3 | 0
Pyrexia (General disorders) | 11 | 5 | 19
Acute sinusitis (Infections and infestations) | 1 | 3 | 0
Cystitis (Infections and infestations) | 1 | 4 | 0
Gastroenteritis (Infections and infestations) | 5 | 2 | 4
Influenza (Infections and infestations) | 8 | 3 | 5
Nasopharyngitis (Infections and infestations) | 2 | 9 | 13
Upper respiratory tract infection (Infections and infestations) | 13 | 6 | 9
Urinary tract infection (Infections and infestations) | 2 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 5
Blood creatine phosphokinase increased (Investigations) | 2 | 2 | 4
Blood glucose increased (Investigations) | 2 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
Dizziness (Nervous system disorders) | 4 | 7 | 6
Migraine (Nervous system disorders) | 6 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03333109/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT03333109/SAP_001.pdf